CLINICAL TRIAL: NCT03359369
Title: Prognostic Value of Serum Cholesterol and Triglyceride in Septic and Non Septic Patients: Randomized Double Blinded Study
Brief Title: Prognostic Value of Serum Cholesterol and Triglyceride in Septic and Non Septic Patients
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, doaa rashwan, assistant professor, Beni-Suef University
Other Study IDs: doaa rashwan
Record Dates: First submitted 2017-11-24; First posted 2017-12-02 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Septic Patients; Nonseptic Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic Patients
  Interventions: Diagnostic Test: level of serum cholesterol and triglyceride
- Non Septic Patients
  Interventions: Diagnostic Test: level of serum cholesterol and triglyceride

INTERVENTIONS:
Diagnostic Test: level of serum cholesterol and triglyceride — other

SUMMARY:
The primary outcome of this study is to evaluate the difference between the level of serum cholesterol and triglyceride in septic and non septic patients in the ICU. .

The secondary outcome will be to find correlation between the level of serum cholesterol and triglyceride and both Acute physiology And Chronic Health Evaluation Score (APACHE) II(19) and quick Sequential Organ Failure Assessment (qSOFA) score (20) and their relation to mortality.

DETAILED DESCRIPTION:
Type and Site of The study:

This study will be be done at Beni-Suef university hospital SICU after approval of the local ethics and research committee and anesthesia department of Beni-Suef University.

DATE AND PERIOD OF THE STUDY:

The study will be done between June 2017 and June 2018

Study population:

The study population will include the patients (age range between 20 and 70)of both sex (septic and non septic patients e.g. trauma patients, post surgical patients) who will be admitted to the surgical intensive care in Beni Suef University hospital.

Sample size estimation:

Sample technique:

The patients will be randomly assigned into two groups, septic patients (groups) according to established consensus definitions (21) or non septic patients (NS) as post surgical and trauma patients.

The following data will be recorded for each patient: age, sex,weight, cause of ICU admission, administration of vasoactive drugs, length of ICU stay, 28-day mortality, administration of vasoactive drugs, days on mechanical ventilation, Acute Physiology and Chronic Health Evaluation II (APACHE II) scores, quick Sequential Organ Failure Assessment (qSOFA) scores will be recorded.

The following laboratory data will be measured:

cholesterol, triglyceride on days 0 (ICU admission), 1, 3, and 7, 10 and 14.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include the patients (age range between 20 and 70) of both sex (septic and non septic patients e.g. trauma patients, post surgical patients) who will be admitted to the surgical intensive care in Beni-Suef University hospital

Exclusion Criteria:

* Age less than 20
* Pregnancy
* ICU readmission
* Dyslipidemia
* Patients with liver disease e.g.hepatitis B,hepatitis C , liver cirrhosis, and hepatocellular carcinoma)
* Concomitant of use immunosuppressive therapy
* Using statin or steroid (≥15mg/day) within the previous 7 days
* Patients who had been treated with corticosteroid therapy for septic shock prior to admission to ICU
* Patients sedated by propofol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include the patients (age range between 20 and 70) of both sex (septic and non septic patients e.g. trauma patients, post surgical patients) who will be admitted to the surgical intensive care in Beni-Suef University hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
change in the level of serum cholesterol and triglyceride | on days 0, 1, 3, and 7, 10 and 14 days
  change in the level of serum cholesterol and triglyceride

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Medicine, Beni-Suef University, Banī Suwayf, Egypt